CLINICAL TRIAL: NCT05707429
Title: Sexual Function and Quality of Life Among Patients Suffering From Inflammatory Bowel Disease During Remmsion
Brief Title: Sexual Function and Quality of Life Among Patients Suffering From Inflammatory Bowel Disease(Inactive Stage)
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Bahaa osman taha, assistant lecturer, Assiut University
Other Study IDs: assiut IBD
Record Dates: First submitted 2023-01-14; First posted 2023-02-01 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Sexual Function Disturbances; Inflammatory Bowel Diseases
MeSH Terms: conditions — Sexual Dysfunctions, Psychological; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy control group: will include patient's relatives or volunteers, who accept to participate in the study through invitation or posters which send or spread it to all staff hospitals about importance of the study.
  Interventions: Other: The Arabic version of The International Index of Erectile Function (IIEF-5); Other: The Sexual Quality of Life Questionnaire Male/Female (SQoL M/F); Other: Assessment of depression and anxiety; Other: The Fatigue assessment scale (16); Other: • Quality of life assessment; Other: The Female Sexual Function Index (FSFI)
- IBD patients inactive group: IBD patients group: they will be recruited from outpatient clinic and inpatient with CD or UC at the Gastroenterology department at Alrajhi hospital.
  CD patients will be assessed by the Crohn's Disease Activity Index a score of less than 150 corresponds to relative disease quiescence (remission); 150 to 219, mildly active disease; 220 to 450, moderately active disease; and greater than 450, severe disease (9).
  Interventions: Other: The Arabic version of The International Index of Erectile Function (IIEF-5); Other: The Sexual Quality of Life Questionnaire Male/Female (SQoL M/F); Other: Assessment of depression and anxiety; Other: The Fatigue assessment scale (16); Other: • Quality of life assessment; Other: The Female Sexual Function Index (FSFI)

INTERVENTIONS:
Other: The Arabic version of The International Index of Erectile Function (IIEF-5) — The Arabic version of The International Index of Erectile Function A self-administered questionnaire that assesses 5 dimensions of sexual function over the most recent 4 weeks. It consists of five questions, including vaginal penetration, maintenance of erection, completion of intercourse, sexual satisfaction, and self-confidence of the patient's sexual arousal and maintenance of an erection. A total score of < 22 is defined as ED .
Other: The Sexual Quality of Life Questionnaire Male/Female (SQoL M/F) — was developed by Symonds et al.,(14) which assesses subjects' feelings toward their sexuality (ranging from 0% to 100%, with higher scores indicating higher SQoL). The SQoL M/F was developed as a condition-specific QoL questionnaire to test the relationship between sexual symptoms and other aspects of general health and sexual QoL.
Other: Assessment of depression and anxiety — Arabic version of Hamilton depression and anxiety rating scale (15): used to measure the severity of anxiety and depressive symptoms, and is widely used in both clinical and research settings.
Other: The Fatigue assessment scale (16) — It is a 10-item self-report scale evaluating symptoms of fatigue. The FAS treats fatigue as a unidimensional construct and does not separate its measurement into different factors. However, in order to ensure that the scale evaluates all aspects of fatigue, it measures both physical and mental symptoms. The total score ranges from 10 to 50, with a higher score indicating more severe fatigue.
Other: • Quality of life assessment — Health related quality of life (HRQoL measure): using the Short Inflammatory Bowel Disease Questionnaire (SIBDQ) (17), which assesses physical, social, and emotional domains of IBD patients' lives (scores range from 10-70, with higher scores indicating better HRQoL) The SIBDQ reflects relevant clinical changes in both CD and UC.
Other: The Female Sexual Function Index (FSFI) — The FSFI includes such parameters as desire, arousal, lubrication, orgasm, satisfaction, and pain. The optimal cutoff score of the FSFI is 26.55, which means that a score at or below this value is defined as female SD.

SUMMARY:
Sexual dysfunction [SD] is a significant health burden characterized by a disturbance in sexual desire and psychophysiological changes in the sexual response cycle, resulting in marked distress and interpersonal difficulty (4). As known, both SD and depression are interrelated, so, depression may be an important determinant of sexual functioning in patients with IBD(5).

DETAILED DESCRIPTION:
Inflammatory Bowel Diseases (IBD), Crohn's disease (CD) and ulcerative colitis (UC), are characterized by a chronically relapsing course (1).

IBD is likely to have a substantial impact on body image, intimacy and sexuality, Because of symptoms like abdominal pain, fatigue, bloating, gas, and diarrhea (2).

Complications may include perianal disease, fistulae and abscesses. Surgery is frequently necessary, sometimes including the placement of a stoma or pouch. Furthermore, mood disorders, mainly depression, are reported to be common in IBD (3) .

Sexual dysfunction [SD] is a significant health burden characterized by a disturbance in sexual desire and psychophysiological changes in the sexual response cycle, resulting in marked distress and interpersonal difficulty (4). As known, both SD and depression are interrelated, so, depression may be an important determinant of sexual functioning in patients with IBD(5).

For female IBD patients, SD mainly manifests as decreased sexual desire, orgasm, and sexual arousal disorder, while for men, the most common symptom is erectile dysfunction (ED) (6).

Friedman and Knowles et al. reported that the prevalence of SD in male and female IBD patients ranged from 44% to 53.9% and 40% to 66%, respectively (7).

However, SD in IBD patients still has not attracted widespread attention, and relevant research studies are scarce.

The current study aims to assess sexual functions in patients with inactive IBD and its associated factors with sociodemographic and clinical characteristics.

assessment sexual function among inflammatory bowel disease during disease inactivity

it will evaluate the predictors and impact of SD on quality of life among those patients

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years old.
* Both sexes
* A stable sexual partner for ≥3 months
* ability to fill in and understand the questionnaire
* sign informed consent and participate voluntarily. For control group: An age-matched control group of healthy men and women, in the same region will also be invited to participate. The controls will eligible if they are 18-50 years of age, have a stable heterosexual relationship for at least 3 months and do not have bowel like IBD or irritable bowel syndrome or psychiatric problems.

Exclusion Criteria:

* Those who couldn't understand or fill out the questionnaire themselves and/or those with mental disorders
* Diagnosis of SD before an IBD diagnosis
* SD compounded by other diseases: cardiovascular and cerebrovascular diseases, lung diseases, liver and kidney dysfunction, diabetic neuropathy, other psychiatric disorders (e.g. depression), and neoplastic diseases, etc.
* History or current use of psychotropic drugs or medications have sexual side effects.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Will include 2 groups: IBD patients inactive group and healthy control group. IBD patients group: they will be recruited from outpatient clinic and inpatient with CD or UC at the Gastroenterology department at Alrajhi hospital.
  Healthy control group: will include patient's relatives or volunteers, who accept to participate in the study through invitation or posters which send or spread it to all staff hospitals about importance of the study.
  All participants will subject to
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
inactive IBD &sexual function of both males | 3 months
  using questionnaire IIEF-5 score It consists of five questions, including vaginal penetration, maintenance of erection, completion of intercourse, sexual satisfaction, and self-confidence of the patient's sexual arousal and maintenance of an erection
  * A total score of < 22 is defined as ED . females using FSFI score.
  * The optimal cutoff score of the FSFI is 26.55, which means that a score at or below this value is defined as female SD

SECONDARY OUTCOMES:
Mean scores for quality of life among inactive IBD patients | 3 months
  (using health related quality of life questionnaire)
  The SQoL M/F was developed as a condition-specific QoL questionnaire to test the relationship between sexual symptoms and other aspects of general health and sexual QoL

CONTACTS AND LOCATIONS:
Overall Officials: ahmed mahmoud abd ella hassan, MD, Study Chair — Assiut university ,andrology departement; mostafa Mohammed Hashem, MD, Study Director — Assiut University; ahmed abdelfadeel maghrapy, MD, Study Director — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt